CLINICAL TRIAL: NCT06549517
Title: Analysis of Efficacy of the Mental Training Tech 245: a Novel Method of Cognitive Stimulation Based on Brain Neuroplastic Ability
Brief Title: Study on the Effectiveness of the MTT24.5 Cognitive Training Program on Cognitive Skills, Brain Volume, and Activation
Acronym: MTT245Cog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Biomedical Research, CONICET (Other)
Responsible Party: Principal Investigator, Carol Kotliar, Chief Clinical Research Laboratory, Institute for Biomedical Research, CONICET
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTT245Cog
Record Dates: First submitted 2024-08-03; First posted 2024-08-12 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Dysfunction
Keywords: ageing; cognitive dysfunction; cerebral neuroplasticiy
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Multisite, prospective, and open-label study involving two arms. Subjects from the general adult population were randomly assigned to either a cognitive intervention group or a no-intervention control group. The intervention consisted of in-person cognitive training over 12 weeks, with baseline and final cognitive evaluations. A sub-study will investigate neuroimaging changes in brain volume and activation as parameters of neuroplasticity stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group-MTT24.5 (Active Comparator): Subjects are assigned to 12 cognitive training in-person sessions of the MTT245 program by a validated trainer. Cognitive evaluations are made initially week 1 and at the end of the intervention at week 12.
  Interventions: Behavioral: Cognitive training
- Control group (No Intervention): Subjects are assigned to a controlled arm whereas no intervention were done. They should underwent the same cognitive evaluations than active comparator at week 1 and 12.

INTERVENTIONS:
Behavioral: Cognitive training — MTT24.5 consists in the learning of 40 new datas or knowledges, along 24.5 hours distributted on classes or sessions, during which an average of 3.5 new pieces of knowledge are taught and reinforced through training. Participants are trained using 4 techniques assigned to each new piece of information from a total of 100 available techniques. These techniques include the use of non-dominant skills, literacy in Braille for sighted individuals, and performing 5 actions simultaneously. Each technique is designed to aid in the memorization and learning of new knowledge
  Other Names: Mental Training Tech 245
  Arms: Intervention group-MTT24.5

SUMMARY:
The goal of this study is to evaluate the effectiveness of a cognitive training program called Mental Training Tech 24.5 (MTT24.5). The program aims to enhance brain function and neuronal plasticity in adults who do not have any clinical cognitive impairment. This study will help determine if MTT24.5 improves cognitive abilities and affects brain volume and activation.

The Main Questions it aims to answer are:

Does MTT24.5 improve overall cognitive performance and specific areas like memory, attention, and language skills? What effects does MTT24.5 have on brain volume and activation? How well do participants follow the program, and what are their response patterns?

Study Design

* Researchers will compare the results of participation in the MTT24.5 training versus a control group with no intervention. Participants will be randomly assigned to either the MTT24.5 program or the control group.
* The study involves adults aged 30 and older from the general population who do not have clinical cognitive impairment.
* The intervention includes attending 12 weekly in-person sessions, each lasting about 2 hours, for a total of 24.5 hours.
* The study will assess cognitive performance, brain volume, and activation, as well as monitor adherence to the program and response patterns.

Participants will:

* Engage in the MTT24.5 program or the control condition as assigned.
* Complete cognitive assessments to measure performance in various domains.
* Undergo brain imaging to evaluate changes in brain volume and activation.

DETAILED DESCRIPTION:
Neuronal plasticity presents a promising approach to addressing a pressing contemporary challenge: the intersection of increased life expectancy with the risks of cognitive decline, dementia, and loss of independence. A wealth of literature highlights the potential of various neuronal plasticity stimulation strategies in bolstering cognitive abilities. However, while much focus has been dedicated to using these techniques for neurological rehabilitation, there remains a paucity of evidence regarding their efficacy in maintaining and enhancing cognitive functions in the generally healthy population. In line with this, the cognitive training protocol 'Mental Training Tech 24.5' (MTT24.5) is grounded in the principles of neuronal plasticity and aims to improve cognitive development. It specifically focuses on enhancing memory, reasoning speed, and attention in adults through a conceptual model that posits explicit learning as a direct stimulus for neuronal plasticity.

II) AIMS:

Primary Objectives:

Evaluate the effects of MTT24.5 on cognitive abilities such as memory, attention, orientation, verbal fluency, language, and visuospatial skills.

Assess the effects of MTT24.5 on brain structure and activation, including brain volumes in globally standardized areas and those associated with cognitive abilities, according to cognitive brain areas with taxonomic mapping.

Determine if there are response phenotypes based on individual baseline characteristics, such as age, gender, lifestyle factors, medical history, medications, family history of dementia, diet, and baseline cognitive reserve score.

Secondary Objective:

Analyze the tolerance and adherence to MTT24.5 and its association with outcomes related to cognitive variables, as well as structural and/or functional brain changes.

III) METHODS

Design:

This is a multisite, prospective, randomized open clinical study conducted between March and October 2023.

Regulatory Approvals:

The trial was approved by the review board and the local ethics committee. All participants provided written consent. This study followed the Consolidated Standards of Reporting Trials (CONSORT) reporting guideline.

Evaluations:

* Cognitive Reserve Score (CRS): A validated cognitive reserve scale authorized from Roldan L. et al. The CRS records the frequency of cognitively stimulating activities carried out throughout life. It includes 24 items distributed across four aspects: activities of daily living, education/information, hobbies, and social life. The CRS will be obtained for each subject at baseline (pre-intervention) and after 12 weeks of participation.
* Medical and Lifestyle History Form: A self-administered medical and lifestyle history form called STEPS 5, adapted from www.who.int/chp/steps, and previously used in the Latin American OPTIMO study. This form will be administered to each subject at baseline (pre-intervention).
* The Addenbrooke's Cognitive Examination-III (ACE-III): A brief cognitive test that evaluates five cognitive abilities: attention, memory, verbal fluency, language, and visuospatial skills. The ACE-III score will be obtained for each subject at baseline (pre-intervention) and post-intervention.
* Brain Magnetic Resonance Imaging (BMRI): Brain volume and activation information will be obtained from this study, conducted on a subset of subjects at baseline (pre-intervention) and post-intervention.

Description of the Intervention:

MTT24.5 is a structured program consisting of 40 new pieces of knowledge and 100 learning techniques.developed as a binomial DATA/TECH program, provides the brain with new knowledge (DATA) classified into formal, natural, social, and cultural areas. The TECH consists of 100 high-impact cognitive stimulation modalities designed to enhance memory, attention, verbal fluency, and visuospatial skills. Techniques include methods such as learning to read the information in Braille, writing it with the non-dominant hand, or reinforcing the concept across various domains simultaneously. Each piece of new information and technique is codified and identified with a number throughout the protocol. This integration is intended to promotes changes in brain functionality, improves synaptic efficiency, and achieves permanent plastic changes. The program spans approximately 24.5 hours over 12 weeks, comprising weekly in-person training sessions of 1.5 hours each, supplemented by an additional average of 4 hours of weekly online activities.

The data or new knowledges were selected through an extensive search of relevant knowledge from the basic sciences (natural, cultural, formal, and social sciences). To be included, the data should be expressible in a concise concept stated in a maximum of 15 words, around which an explanation is built using visual animation and emotional aspects or experiential learning during a 10-minute session. The second part of the session aims to promote the integration of the new knowledge into an individual's cognitive reserve, employing cognitive TECHS, which consist of exercises designed for this purpose. TECHS selection was based on a review of peer-reviewed articles demonstrating the effectiveness of cognitive training in improving specific cognitive abilities investigated in the study. We identified 25 cognitive training studies with appropriate tools published between 2000 and 2022. The possible combinations of these tools yielded 75 possibilities regarding the association between 2 to 5 techniques for learning the same data, indicating either consecutive or simultaneous actions.

24.5 represents the total hours assigned to the program duration, based on similar training distributions reported in the ACTIVE TRIAL (The Advanced Cognitive Training for Independent and Vital Elderly).

Detailed descriptions of the statistical analysis plan can be found in the attached document, SA

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 years and above.
* Ability to understand instructions for the training tasks.
* Addenbrooke Cognitive Examination score >70.

Exclusion Criteria:

* Planned absences that would hinder participation in the program.
* Hearing, visual, or motor deficits that would impede participation in the program.
* History of severe degenerative neurological diseases, as these conditions may significantly impact brain plasticity and cognitive abilities.
* History of severe psychiatric disorders, as they may influence brain reorganization and complicate the interpretation of results.
* Unstable treatment or planned changes in medication that may affect brain function and alter results.
* History of current or recent excessive substance use (within the past 6 months), including alcohol or drugs, as these substances may influence brain function and neuroplasticity.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Global Cognitive Ability | immediately after the intervention
  The primary study outcome, cognitive ability changes, was assessed through the difference between the post intervention Addenbrooke's Cognitive Examination III (ACE) score and the pre intervention ACE score. This score ranges from 0 to 100. he ACE Score ranges from 0 to 100. A value less than 85 es considered as cognitive moderate impairment.

SECONDARY OUTCOMES:
Change in memory, and /or attention, and/or verbal fluency, and/or language, and/or visuospatial skills abilities. | immediately after the intervention
  Each ability outcome was assessed using the respective sub-dimensions of the ACE score and computing the difference between post intervention and pre intervention sub-score:
  * Memory ability sub-score
  * Attention ability sub-score
  * Orientation ability sub-score
  * Verbal fluency ability sub-score
  * Language ability sub-score
  * Visuospatial skills ability sub-score The memory ability sub-score ranges from 0 to 26, the attention abilities sub-score ranges from 0 to 8, the attention abilities sub-score ranges from 0 to 10, the verbal fluency sub-score ranges from 0 to 14, the language sub-score ranges from 0 to 16, and the visuospatial skills abilities sub-score ranges
Rate of Adherence | immediately after the intervention
  Adherence or compliance with the study protocol was assessed through the number of days that participant completed ("on site days"); as participants were instructed and reminded to complete weekly sessions, the number of active days was used as the primary measure of a participant's ongoing engagement and compliance with the study protocol.
Change in Brain Volume and Activation | immediately after the intervention
  Changes are reported as the volumes and/or activation obtained values of different structures of the brain, both in absolute terms (cm3) and relative (% of the total), and values reference of normal populations corrected for age and sex.

CONTACTS AND LOCATIONS:
Overall Officials: Carol V Kotliar, PhD, Principal Investigator — BIO; Carol V Kotliar, PhD, Principal Investigator — Institute for Biomedical Research, CONICET
Locations (1):
- Espacio Santa Maria, San Isidro, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
At the time of publication, and upon aproval of the request by a scientific board, all IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At the time of publication in a peer review journal
Access Criteria: By written request to the PI, accompanied by a letter explaining objectives of the IPD to be shared and research group institution or antecedents of the individual if not an institution.
URL: http://espaciosantamaria.com.ar

REFERENCES:
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Lindenberger U. Human cognitive aging: corriger la fortune? Science. 2014 Oct 31;346(6209):572-8. doi: 10.1126/science.1254403. PMID 25359964
- [Background] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Background] Snowdon DA; Nun Study. Healthy aging and dementia: findings from the Nun Study. Ann Intern Med. 2003 Sep 2;139(5 Pt 2):450-4. doi: 10.7326/0003-4819-139-5_part_2-200309021-00014. PMID 12965975
- [Background] Rebok GW, Ball K, Guey LT, Jones RN, Kim HY, King JW, Marsiske M, Morris JN, Tennstedt SL, Unverzagt FW, Willis SL; ACTIVE Study Group. Ten-year effects of the advanced cognitive training for independent and vital elderly cognitive training trial on cognition and everyday functioning in older adults. J Am Geriatr Soc. 2014 Jan;62(1):16-24. doi: 10.1111/jgs.12607. Epub 2014 Jan 13. PMID 24417410
- [Background] Feingold A. New Approaches for Estimation of Effect Sizes and their Confidence Intervals for Treatment Effects from Randomized Controlled Trials. Quant Method Psychol. 2019;15(2):96-111. doi: 10.20982/tqmp.15.2.p096. PMID 32775313
- [Background] Masic V, Secic A, Trost Bobic T, Femec L. Neuroplasticity and Braille reading. Acta Clin Croat. 2020 Mar;59(1):147-153. doi: 10.20471/acc.2020.59.01.18. PMID 32724286
- [Derived] Kotliar C, Olmos L, Koretzky M, Jauregui R, Delia T, Cingolani O. A new program for systematically enhancing cognitive reserve in healthy adults: A pilot randomized active-controlled clinical trial. PLoS One. 2025 Oct 1;20(10):e0331193. doi: 10.1371/journal.pone.0331193. eCollection 2025. PMID 41032503

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT06549517/SAP_000.pdf